CLINICAL TRIAL: NCT01277341
Title: Safety and Efficacy of Bepotastine Besilate Nasal Spray in the Treatment of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S00082
Record Dates: First submitted 2011-01-07; First posted 2011-01-14 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2% Twice a day (Experimental): Bepotastine Besilate Nasal Spray 2% Twice a day
  Interventions: Drug: Bepotastine Besilate Nasal Spray 2% Twice a day
- 3% Twice a day (Experimental): Bepotastine Besilate Nasal Spray 3% Twice a day
  Interventions: Drug: Bepotastine Besilate Nasal Spray 3% Twice a day
- 4% Twice a day (Experimental): Bepotastine Besilate Nasal Spray 4% Twice a day
  Interventions: Drug: Bepotastine Besilate Nasal Spray 4% Twice a day
- Placebo (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: Bepotastine Besilate Nasal Spray 2% Twice a day — nasal spray
  Arms: 2% Twice a day
Drug: Bepotastine Besilate Nasal Spray 3% Twice a day — nasal spray
  Arms: 3% Twice a day
Drug: Bepotastine Besilate Nasal Spray 4% Twice a day — nasal spray
  Arms: 4% Twice a day
Drug: Placebo Nasal Spray — nasal spray
  Arms: Placebo

SUMMARY:
This is an efficacy study of bepotastine besilate nasal spray in seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 12 years of age with a history of mountain cedar allergy

Exclusion Criteria:

* No active nasal infection or nasal abnormality that would affect subject safety or symptom assessments

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2% Twice a Day | 3% Twice a Day | 4% Twice a Day | Placebo
Started | 150 | 150 | 149 | 152
Completed | 146 | 145 | 145 | 146
Not Completed | 4 | 5 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% Twice a Day | 3% Twice a Day | 4% Twice a Day | Placebo | Total
Number analyzed (Participants) | 150 | 150 | 149 | 152 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (15.2) | 40.9 (15.6) | 41.6 (15.9) | 39.5 (14.9) | 40.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 94 | 87 | 90 | 363
  Male | 58 | 56 | 62 | 62 | 238

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Pre-Dose) in Subject-rated Reflective TNSS
Description: Total nasal symptom score (TNSS) was the summed scores for nasal pruritus [itching], rhinorrhea [runny nose], nasal congestion, and sneezing. Individual nasal symptoms were each rated on a 4-point scale from 0-3 (0=Absent, 1=Mild, 2=Moderate, 3=Severe), with no half-unit assessments. TNSS was the sum score of 4 nasal symptoms with a minimum score of 0 units and a maximum score of 12 units, with higher score corresponding to increased nasal allergy symptoms. Morning and evening scores were averaged.
Time Frame: Baseline, 14 days
Population: All randomized participants were included in the analysis population, with no imputation of missing data at 14 days.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2% Twice a Day | 3% Twice a Day | 4% Twice a Day | Placebo
Number analyzed (Participants) | 135 | 134 | 128 | 130
score on a scale | -1.84 (1.80) | -1.71 (1.97) | -1.47 (1.88) | -0.99 (1.69)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | 2% Twice a Day | 3% Twice a Day | 4% Twice a Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/150 | 1/150 | 0/149 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/150 | 1/150 | 0/149 | 0/152
Other Adverse Events (participants affected / at risk) | 25/150 | 22/150 | 22/149 | 10/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2% Twice a Day (N=150) | 3% Twice a Day (N=150) | 4% Twice a Day (N=149) | Placebo (N=152)
Death (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2% Twice a Day (N=150) | 3% Twice a Day (N=150) | 4% Twice a Day (N=149) | Placebo (N=152)
Mild taste following instillation (General disorders) | 25 (150) | 22 (150) | 22 (149) | 10 (152)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor directly for details.